CLINICAL TRIAL: NCT04062591
Title: Efficacy of Piroxicam as a Perioperative Analgesic for Patients Undergoing Fixation of Maxillofacial Fractures
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, Associate professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 54/ 2018
Record Dates: First submitted 2019-08-17; First posted 2019-08-20 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Pain
Keywords: piroxicam; VAS; fractures
MeSH Terms: conditions — Pain, Postoperative; Fractures, Bone | interventions — Piroxicam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- piroxicam (Active Comparator): piroxicam group who received induction with piroxicam(0.4mg/kg) IM
  Interventions: Drug: Piroxicam group
- placebo (Sham Comparator): saline IM in the same dose of piroxicam
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Piroxicam group — patients will receive 0.4 mg/kg piroxicam IM
  Other Names: piroxicam
  Arms: piroxicam
Drug: Placebo — saline IM in the same dose of piroxicam
  Arms: placebo

SUMMARY:
At Eldemerdash Hospital at Ain Shams University in Egypt, 72 adult patients (16 to 25 years old) who had mandibular or maxillary fractures were treated with open reduction and internal stabilization. Patients were divided into two categories. (31 patients each) Using randomly generated data from computer, the piroxicam group received 0.4 mg/kg of intramuscular piroxicam, while the general anesthesia group (GA group) did not receive piroxicam.

The overall amount of rescue analgesic dosage and postoperative complications like nausea and vomiting were therefore included in the outcomes measurement.

DETAILED DESCRIPTION:
Patients were divided into two groups at random using a computer-generated list: the GA group received no piroxicam and the piroxicam group got a 0.4 mg/kg IM piroxicam induction. Both groups got IV paracetamol (24 mg/kg slowly administered over 20 minutes).

Fentanyl 2 micrograms/kg was administered after general anesthesia was induced and venous access was established. A suitable size endotracheal tube was then placed intranasal, and intubation was aided by Atracurium (0.5 mg/kg). Throughout the operation, 1 MAC isoflurane in a mixture of 50% air and oxygen was used to maintain anesthesia in all patients who were mechanically ventilated in pressure-controlled mode with targeted EtCO2 (30-35 mmHg). An oral pack was also introduced.

After the operation general anesthesia was stopped and the endotracheal tube was removed, Neostigmine 50 mg/kg and atropine sulfate 15 mg/kg were used to reverse muscle relaxation. Patient transportation was made to the post-anesthesia care unit (PACU). Postoperative analgesia was evaluated by a blind investigator using 10 cm- visual analogue scale score which had been explained to the patient on the preoperative visit where: 0 = no pain, 10 = worst possible pain) in the PACU then at 3, 6, 12, 24 hours, if the pain score >3, pethidine 25 mg intravenously and Ondansetron 0.1mg/kg was used for cases with nausea or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 16-25 years old
* ASAI II
* scheduled for open reduction and internal fixation of mandibular or maxillary fractures

Exclusion Criteria:

* a history of convulsion,
* gastrodudenal ulcer
* hematological disorders
* patient suffering from hepatic or renal dysfunction
* concomitant use of anticoagulants
* refusal of the patients to participate
* patients younger than 12 years

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
rescue dose of analgesic | 24 hours
  patients needed additional doses of rescue analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Effat, professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams U, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol statistical analysis data analysis
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 7 months
Access Criteria: Data were analyzed using SPSS Statistics version 23 (IBM© Corp., Armonk, NY, USA). Normally distributed numerical data were presented as mean and SD, and skewed data were presented as median and interquartile range. Qualitative data were presented as number and percentage or ratio. Normally distributed numerical data were compared using the unpaired t-test. Skewed numerical data were compared using the Mann-Whitney test and categorical data were compared using Fisher's exact test.